CLINICAL TRIAL: NCT00245141
Title: Phase II Trial of Short VAC1.2 Therapy for Low-Risk A Group Patients With Rhabdomyosarcoma
Brief Title: Vincristine, Dactinomycin, and Cyclophosphamide With or Without Radiation Therapy in Treating Patients With Embryonal Rhabdomyosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Japan Rhabdomyosarcoma Study Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: JRSG-UHA-PED03-01; CDR0000453316 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Sarcoma
Keywords: embryonal childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Dactinomycin; Cyclophosphamide; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: dactinomycin
Drug: cyclophosphamide
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vincristine, dactinomycin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells. Giving more than one drug (combination chemotherapy) with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vincristine, dactinomycin, and cyclophosphamide together with or without radiation therapy works in treating patients with embryonal rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free survival rate in patients with low-risk embryonal rhadomyosarcoma treated with a shortened treatment schedule of vincristine, dactinomycin, and cyclophosphamide with or without radiotherapy.

OUTLINE: Patients receive vincristine IV, dactinomycin IV, and cyclophosphamide IV. Patients may also undergo radiotherapy. Treatment repeats every 3 weeks for up to 8 courses (total of 24 weeks) in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of embryonal rhabdomyosarcoma

  * Primary operation for pathological diagnosis within the past 42 days
  * The following variants are eligible:

    * Botryoid
    * Spindle cell
    * Anaplastic
* Meets 1 of the following stage criteria:

  * Stage I, clinical group I or II (N0), defined by all of the following criteria:

    * Favorable site, including orbit, head, and neck (excluding parameningeal sites), genitourinary region (excluding bladder/prostate sites), or biliary tract
    * Tumor any size
    * Completely resected disease OR microscopic residual disease
    * Lymph nodes clinically negative
  * Stage I, clinical group III (N0), defined by all of the following criteria:

    * Favorable site
    * Tumor any size
    * Gross residual disease allowed (orbit only)
    * Lymph nodes clinically negative
  * Stage II, clinical group I (N0, Nx), defined by all of the following criteria:

    * Unfavorable site (any sites not listed as favorable sites)
    * Tumor ≤ 5 cm in diameter
    * Completely resected disease
    * Lymph nodes clinically negative OR lymph node involvement unknown

PATIENT CHARACTERISTICS:

Performance status

* 0-3

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 7.5 g/dL

Hepatic

* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.5 times ULN
* Bile acid ≤ 2.5 times ULN

Renal

* Creatinine based on age as follows:

  * < 0.8 mg/dL (for patients < 5 years of age)
  * < 1.2 mg/dL (for patients 5-9 years of age)
  * < 1.5 mg/dL (for patients ≥ 10 years of age)

Cardiovascular

* No severe heart disease

Other

* Not pregnant or nursing
* Must have acceptable organ function for age
* No uncontrolled infection
* No other active malignancy
* No other treated malignancy within the past 5 years
* No hypersensitivity to study drugs
* No Charcot-Marie-Tooth disease
* No chickenpox

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior anticancer chemotherapy

Endocrine therapy

* Prior anticancer steroids allowed

Radiotherapy

* No prior radiotherapy

Other

* No concurrent pentostatin

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2004-05; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival as measured by Kaplan-Meier method 3 years after study entry

SECONDARY OUTCOMES:
Overall survival as measured by Kaplan-Meier method 3 years after study entry
Progression-free survival as measured by Kaplan-Meier method during events
Complete response rate (orbit, group III only) at completion of study treatment
Rate of toxicity as measured by NCI-CTC v 2.0 3 years after study entry

CONTACTS AND LOCATIONS:
Overall Officials: Hajime Hosoi, Study Chair — Kyoto Prefectural University of Medicine; Masa-aki Kumagai, MD — National Center for Child Health and Development
Locations (51):
- Japan (51):
  - Anjo Kosei Hosptial, Anjo, Aichi-ken
  - Aichi Medical University, Nagakuti, Aichi-ken
  - National Hospital Orgnization Nagoya Medical Center, Nagoya, Aichi-ken
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - National Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kurume University School of Medicine, Kurume, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu Municipal Hospital, Gifu, Gifu
  - Gifu University Graduate School of Medicine, Gifu, Gifu
  - Gunma Children's Medical Center, Seta-gun, Gunma
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization - Medical Center of Kure, Kure, Hiroshima
  - Sapporo Medical University, Sapporo, Hokkaido
  - Hokkaido University Graduate School of Medicine, Sapporo, Hokkaido
  - Kobe City General Hospital, Kobe, Hyōgo
  - Ibaraki Children's Hospital, Mito, Ibaraki
  - University of Tsukuba, Tsukuba, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical University, Kanazawa, Ishikawa-ken
  - Kagoshima University, Kagoshima, Kagoshima-ken
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - National Center for Child Health and Development, Tokyo, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Yokohama City University, Yokohama, Kanagawa
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Miyazaki Medical College University of Miyazaki, Miyazaki-gun, Miyazaki
  - Nagano Children's Hospital, Toyoshina-machi, Nagano
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Osaka City University, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka City General Hospital, Suita-shi, Osaka
  - Osaka University Graduate School of Medicine, Suita-shi, Osaka
  - Osaka Medical College, Takatsuki, Osaka
  - Dokkyo University School of Medicine, Koshigaya, Saitama
  - Saitama Children's Medical Center, Saitama, Saitama
  - National Defense Medical College, Tokorozawa, Saitama
  - Shiga University of Medical Science, Ōtsu, Shiga
  - Shimane Prefectural Central Hospital, Izumo, Shimane
  - Shimane University Hospital, Izumo, Shimane
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Tokyo Metropolitan Kiyose Children's Hospital, Kiyosei, Tokyo
  - National Cancer Center Hospital, Tokyo, Tokyo
  - St. Luke's International Hospital, Tokyo, Tokyo
  - Tokyo Medical and Dental University, Tokyo, Tokyo
  - Toho University School of Medicine, Tokyo, Tokyo
  - Keio University School of Medicine, Tokyo, Tokyo
  - Nihon University Itabashi Hospital, Tokyo, Tokyo
  - Toyama University Hospital, Toyama, Toyama
  - Yamagata University Hospital, Yamagata, Yamagata
  - Hokkaido Medical Center for Child Health and Rehabilitation, Sapporo